CLINICAL TRIAL: NCT02494687
Title: Domperidone Expanded Access Program for Oncology Patients With Gastroparesis Who Have Failed Standard Therapy
Status: Available | Type: Expanded Access
Sponsor: Eastern Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: EP2014022
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Oncology Patients With Gastroparesis
MeSH Terms: interventions — Domperidone

INTERVENTIONS:
Drug: Oral Domperidone — 10 mg of oral domperidone administered (four times a day) for two weeks
Drug: Oral Domperidone — Increased to 20 mg four times a day for 2 weeks at the Investigator's discretion
Drug: Oral Domperidone — Increased to 30 mg four times a day at the Investigator's discretion

SUMMARY:
Gastroparesis is a digestive disorder in which motility of the stomach is either slowed or absent. The gastroparesis prevents normal digestion from occurring. The purpose of this study is to provide oral Domperidone offered under the U.S. Food and Drug Administration (FDA) expanded access program, to patients that, based on the treating doctor's assessment, could benefit from , a prokinetic effect for the relief of refractory gastroesophageal reflux disease with upper gastrointestinal (GI) symptoms, gastroparesis, and chronic constipation.

DETAILED DESCRIPTION:
At the discretion of the Investigator, 10-30 mg of oral domperidone is administered QID (four times a day). The Investigator will be starting patients on 10 mg four times a day for 2 weeks, then increase to 20 mg four times a day for 2 weeks. The participant will be evaluated at each time point. If the participant still is not having relief of symptoms the investigator may increase their dose to 30mg four times a day.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18 and older
3. Symptoms or manifestations secondary to GERD (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms), gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation refractory to standard therapy.
4. Patients must have a comprehensive evaluation (physical exam and also may include EGD, gastric emptying study, as clinically necessary) to eliminate other causes of their symptoms.
5. Patient has signed informed consent for the administration of domperidone that informs the patient of potential adverse events including:

   * increased prolactin levels
   * extrapyramidal side-effects
   * breast changes
   * cardiac arrhythmias including QT prolongation and death

Exclusion Criteria:

History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Patients with minor forms of ectopy (PACs) are not necessarily excluded.

1. Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QTc (QTc> 450 milliseconds for males, QTc>470 milliseconds for females).
2. Clinically significant electrolyte disorders.
3. Gastrointestinal hemorrhage or obstruction
4. Presence of a prolactinoma (prolactin-releasing pituitary tumor).
5. Pregnant or breast feeding female
6. Known allergy to domperidone

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Regional Medical Center, Inc., Philadelphia, Pennsylvania, United States